CLINICAL TRIAL: NCT05825495
Title: Postoperative Pain Management on Uvulopalatopharyngoplasty Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Li-Jen Hsin (Other)
Responsible Party: Sponsor-Investigator, Li-Jen Hsin, Principal Investigator, Chang Gung Memorial Hospital
Organization: Chang Gung Memorial Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202202344A3
Record Dates: First submitted 2023-04-11; First posted 2023-04-24 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Pain, Postoperative; Obstructive Sleep Apnea-hypopnea Syndrome; Pain, Acute
Keywords: dinalbuphine sebacte; nalbuphine; Naldebain; Uvulopalatopharyngoplasty
MeSH Terms: conditions — Pain, Postoperative; Acute Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Active Comparator): Subjects will intragluteally injected with a dose of 150 mg dinalbuphine sebacate at least 12 hours before surgery. During intra- and post-operative period, the pain management will execute following our routine practice.
  Interventions: Drug: Dinalbuphine sebacate; Other: Routine practice
- Control group (Sham Comparator): The pain management will peri-operatively execute following our routine practice without dinalbuphine sebacate administration.
  Interventions: Other: Routine practice

INTERVENTIONS:
Drug: Dinalbuphine sebacate — A single dose of 150 mg dinalbuphine sebacate will be intragluteally administrated at least 12 hours before surgery.
  Other Names: Naldebain
  Arms: Experimental group
Other: Routine practice — Within 3 days after surgery, paracoxib will be administrated twice a day. Ketorolac will intravenously give once breakthrough pain occurring. Enteral acetaminophen will be take regularly within 14 days after surgery.

SUMMARY:
This is a randomized controlled study, aimed to investigate the effects of dinalbuphine sebacate (DS) on patients having uvulopalatopharyngoplasty (UPPP). DS is a prodrug of nalbuphine, a mixed agonist-antagonist opioid. The mean absorption time for the complete release of DS into systemic circulation is approximately 145 h, which could theoretically provide extended analgesic effects for up to 6 days. Patients diagnosed with obstructive sleep apnea are generally associated with higher risks towards opioid side effects, especially respiratory depression. Post-UPPP pain managing should be cautiously arranged and executed. We hypothesize that the combination of our routine practice and DS will improve the outcomes after Uppp.

DETAILED DESCRIPTION:
Within 4 weeks before uvulopalatopharyngoplasty, patients are invited for this study. After written informed consent gained, the eligibilities are checked. Eligible patients are arrogated into experimental or control group randomly prior to surgery. Experimental group receives the DS administration at least 12 hours before surgery. During peri-operative period, pain management are conducted following our routine practice. Pain intensity, consumption of analgesics, adverse events, swallow function and life quality are all assessed and recorded within 14 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

* aged between 20 and 65.
* diagnosed with obstructive sleep apnea.
* arranged to undergo uvulopalatopharyngoplasty.
* classified as ASA I, II, or III.

Exclusion Criteria:

* can not comply with study protocol.
* BMI > 34 kg/m2.
* history of chronic pain.
* history of narcotics or alcohol abuse.
* allergic to NSAID.
* diagnosed as diabetes mellitus with poor glycemic control.
* diagnosed with severe cardiovascular or respiratory diseases.
* judged as an unsuitable subject by investigators.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2024-04-23 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | within 3 days after surgery
  Pain intensity will be assessed via numeric rating scale, 0 means no pain and 10 means the worst pain imaged.

SECONDARY OUTCOMES:
Pain intensity | within 14 days after surgery
  Pain intensity will be assessed via numeric rating scale, 0 means no pain and 10 means the worst pain imaged.
Consumption of analgesics | within 3 days after surgery
  Consumption of analgesics will be summarized by drug categories, routes and the individual days administrated.
Consumption of analgesics | within 14 days after surgery
  Consumption of analgesics will be summarized by drug categories, routes and the individual days administrated.
Percentage of patients consuming analgesics | within 3 days after surgery
  Percentage and number of patients consuming analgesics will be summarized by drug categories, route and the individual days administrated.
Incidence of adverse events | within 3 days after surgery
  Percentage and number of patients suffering from adverse events will be summarized by the individual days.
Incidence of adverse events | within 14 days after surgery
  Percentage and number of patients suffering from adverse events will be summarized by the individual days.
EAT-10 (Eating Assessment Tool) | 1 day, 3 days, 7 days and 14 days after surgery
  EAT-10 is a dysphagia assessment that helps to measure swallowing difficulties. There are 10 questions in the questionnaire. Each question has 5 levels, 0 means no problem and 4 means severe problem.
MD Anderson Dysphagia Inventory | 1 day, 3 days, 7 days and 14 days after surgery
  The MDADI is the first validated and reliable self-administered questionnaire designed specifically for evaluating the impact of dysphagia on the QOL of patients with head and neck cancer. There are 20 questions in the questionnaire. Each question has five levels, including strongly disagree, disagree, no opinion, agree, strongly agree.

CONTACTS AND LOCATIONS:
Overall Officials: Li-Jen Hsin, MD, Principal Investigator — Linkou Chang Gung Hospital